CLINICAL TRIAL: NCT05272059
Title: A Randomized, Investigator and Participant Blinded, Placebo Controlled, Multiple Ascending Dose, Two Part Design Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of MHS552 in Adults With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Multiple Ascending Dose Study of MHS552 in Adults With Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CMHS552B12101
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus, T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: Cohort 1 - MHS552 low dose (Experimental): Participants will receive MHS552 low dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part A: Cohort 1, 2, 3 - Placebo (Placebo Comparator): Participants will receive placebo once weekly subcutaneously for 4 weeks
  Interventions: Drug: Placebo
- Part A: Cohort 2 - MHS552 medium dose (Experimental): Participants will receive MHS552 medium dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part A: Cohort 3 - MHS552 high dose (Experimental): Participants will receive MHS552 high dose once weekly subcutaneously for 4 weeks
  Interventions: Drug: MHS552
- Part B: MHS552 (Experimental): Participants will MHS552 (dose to be determined) once weekly subcutaneously for 12 weeks
  Interventions: Drug: MHS552
- Part B: Placebo (Placebo Comparator): Participants will receive placebo once weekly subcutaneously for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHS552 — MHS552 will be administered once weekly as subcutaneous injection for 4 (Part A) or 12 weeks (Part B)
  Arms: Part A: Cohort 1 - MHS552 low dose; Part A: Cohort 2 - MHS552 medium dose; Part A: Cohort 3 - MHS552 high dose; Part B: MHS552
Drug: Placebo — Placebo will be administered once weekly as subcutaneous injection for 4 (Part A) or 12 weeks (Part B)
  Arms: Part A: Cohort 1, 2, 3 - Placebo; Part B: Placebo

SUMMARY:
The purpose of this two-part multiple ascending dose study is to evaluate the safety and tolerability of multiple doses of MHS552 in adults with type 1 diabetes mellitus. Participants will be treated for 4 or 12 weeks followed by an 8 week follow-up period

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, investigator and participant blinded, placebo controlled, multiple ascending dose (MAD) study in adults with type 1 diabetes mellitus (adults aged 18-45 years, inclusive, diagnosed with T1DM within 5 years at the time of screening). This MAD study will be conducted in two sequential parts, Part A and Part B.

In Part A, after an screening period of up to 28 days, participants will be randomized (in a 3:1 ratio) to MHS552 or placebo administered subcutaneously (s.c.) weekly for four weeks of treatment. Part A will consist of up to 3 cohorts (low, medium, high dose), with approximately 4-8 participants completing each cohort (total of approximately 16 participants). Participants will be followed-up during 8 weeks post last dose. The total duration of study participation of Part A is approximately 106 Days.

In Part B, after a screening period of up to 28 days, approximately 12 participants will be randomized (in a 2:1 ratio) to MHS552 or placebo administered s.c. weekly for 12 weeks of treatment (dose level 4). Participants will be followed-up during 8 weeks post last dose with End of Study (EoS) visit at Day 134. The total duration of study participation of Part B is approximately 162 Days.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ages 18 to 45, inclusive, body weight between ≥40 to ≤150 kg, inclusive, with T1DM, a maximum of 5 years from T1DM diagnosis at screening.
* Evidence of one or more T1DM autoantibody(ies) including glutamic acid decarboxylase (anti GAD), protein tyrosine, phosphatase-like protein (anti-IA-2); zinc transporter 8 (anti-ZnT8); islet cell (cytoplasmic) (anti-ICA)
* Residual pancreatic β-cell function (fasting C-peptide >100 pmol/L [0.30 ng/mL] or random C peptide >200 pmol/L [0.60 ng/mL])

Exclusion Criteria:

* History of hypersensitivity to drugs of similar biological class, IL-2 protein analogues, or immunoglobulin (IgG1) proteins, hypersensitivity to any components of the study drug, or history of severe hypersensitivity reaction or anaphylaxis to biological agents, e.g. human monoclonal antibody.
* Use of other investigational drugs or use of immunosuppressive agents at the time of enrollment, or within 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* Diabetes forms other than autoimmune type 1 such as maturity-onset diabetes of the young (MODY), latent autoimmune diabetes of the adult (LADA), acquired diabetes (secondary to medications or surgery), type 2 diabetes by judgement of the investigator.
* Diabetic ketoacidosis within 2 weeks.
* Polyglandular auto-immune disease, including but not limited to: Addison's disease, pernicious anemia, celiac sprue and psoriasis. Treated, stable Hashimoto's thyroiditis is not exclusionary.
* History of capillary leak syndrome (CLS).
* Ongoing, and up to 2 weeks prior to screening, initiation of medications or change in dose of medications that may affect glucose control (e.g, systemic steroids, thiazides, beta blockers).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | Part A: up to 12 weeks; Part B: up to 20 weeks
  Numbers of participants with AEs and SAEs including vital signs, electrocardiograms (ECG) and laboratory results

SECONDARY OUTCOMES:
Area Under Plasma Concentration-time Curve calculated to the end of a dosing interval (AUCtau) for MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the AUCtau profile following multiple doses of MHS552
Maximum ObservBlood Concentrations (Cmax) for MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the Cmax profile following multiple doses of MHS552
Time to Reach Maximum Blood Concentrations (Tmax) of MHS552 | Part A: up to Day 78; Part B: up to Day 134
  Characterize the Tmax profile following multiple doses of MHS552

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No